CLINICAL TRIAL: NCT06718816
Title: A Long-term Follow-up Study to Evaluate the Safety and Effectivity of AL-001 Ophthalmic Injection in Subjects with Wet Age-related Mecular Degeneration (wAMD)
Brief Title: Long-term Follow-up Study of AL-001 Ophthalmic Injection in Subjects with WAMD
Status: Recruiting | Type: Observational
Sponsor: Beijing Anlong Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AL-001-LT
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Wet Age-related Macular Degeneration (wAMD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The subjects received AL-001 ophthalmic injection: Evaluate long-term safety and efficacy

SUMMARY:
This study is designed to evaluate long-term safety and efficacy of AL-001 ophthalmic injection following suprachoroidal space(SCS) administration in subjects with wAMD. Eligible patients, are those who were previously enrolled in a clinical study in which they received a single dose of AL-001 administered via suprachoroidal space injection.

ELIGIBILITY:
Inclusion Criteria:

* The subjects enrolled in AL-001 study and received AL-001 ophthalmic injection.
* The subject or their legal representative agrees to participate in this study and signs a written ICF.
* The subjects are willing and able to follow planned visits and procedures.

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled in AL-001-01 study and received AL-001 ophthalmic injection.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
AE/SAE | month 48
  Incidence and severity of ophthalmic and systematic AE/SAE.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity(BCVA) | month 48
  Change in BCVA from baseline
The mean and frequency of anti-VEGF injections | month 48
  The mean and frequency of subjects with wAMD receiving anti-VEGF injections

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Hospital, Beijing, Beijing Municipality, China